CLINICAL TRIAL: NCT05620251
Title: Immunogenicity of SARS-CoV-2 BNT162b2 Vaccine in Adolescents With Type 1 Diabetes: A Prospective Observational Study
Brief Title: Response to BNT162b2 Vaccine in Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Hamdi Cihan Emeksiz, associate professor, Istanbul Medeniyet University
Other Study IDs: 2022/0190
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: type1diabetes
Keywords: type 1 diabetes; SARS-CoV-2; immunogenicity; antibody; covid-19; adolescents; vaccine; BNT162b2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 infection-naive adolescents with type 1 diabetes
  Interventions: Diagnostic Test: Blood test
- COVID-19 infection-naive healthy controls
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Assessment of humoral immune response

SUMMARY:
Adolescents with type 1 diabetes may be at increased risk for severe coronavirus disease-2019 (COVID-19) and are therefore prioritized for access to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccination. The pivotal trial that assessed the efficacy of the BNT162b2 vaccine among adolescents demonstrated 100% protection against SARS-CoV-2 infection after a two-dose regimen. However, the research did not include adolescents with type 1 diabetes. In this study, the investigators aimed to assess the humoral immune response of infection-naive adolescents with type 1 diabetes following vaccination with the BNT162b2 vaccine in comparison to that of infection-naive healthy controls and the factors associated with that response.

DETAILED DESCRIPTION:
Having either form of diabetes as a comorbidity has been implicated as a risk factor for severe COVID-19. Therefore, vaccination against COVID-19 has been highly recommended for people with diabetes. However, since diabetes is associated with persistent and profound impairments in both innate and acquired immunity, whether the immune system of people with diabetes will be able to mount an adequate antibody (ab) response following COVID-19 vaccination has remained in question. Some studies have reported that adults with diabetes develop an inadequate immune response to hepatitis B vaccines, whereas less consistent results have been reported for varicella-zoster and influenza vaccines. Likewise, certain pediatric studies have found that serum ab titers against hepatitis B surface antigen and pneumococcal antigens were lower in children with type 1 diabetes than in controls following hepatitis B vaccine and unconjugated pneumococcal polysaccharide vaccine administration. In this context, concerns about the effectiveness of COVID-19 vaccines in people with diabetes have led to the investigation of their immunogenicity after vaccination against COVID-19.

Thus far, few studies have explored the ab response of people with diabetes following COVID-19 vaccination. In the majority of studies conducted, the seroconversion rates of people with diabetes were found to be lower than those of age-matched healthy controls. Nonetheless, the majority of the diabetic people included in these studies were still able to elicit a strong ab response. However, most of these studies only enrolled adults with type 2 diabetes. The ab response to COVID-19 vaccination in a pediatric cohort with type 1 diabetes has not been investigated. Thus, in this single-centered prospective observational study, the investigators aimed to analyze the ab response to a widely used and effective mRNA (messenger ribonucleic acid)-based SARS-CoV-2 vaccine, BNT162b2, in adolescents with type 1 diabetes compared to that of healthy controls and the factors associated with that response.

ELIGIBILITY:
Inclusion Criteria for adolescents with type 1 diabetes:

* aged between 12-18 years
* history of diabetes
* willingness to provide informed consent

Exclusion Criteria for adolescents with type 1 diabetes:

* age < 12 years and age > 18 years
* history of chronic disease
* previous episode of COVID-19
* respiratory symptoms up to 14 days before the study
* history of systematic treatment with corticosteroids and/or immunosuppressant medications

Inclusion Criteria for controls:

* aged between 12-18 years
* good health
* no previous history of diabetes
* willingness to provide informed consent

Exclusion Criteria for controls:

* age < 12 years and age > 18 years
* history of chronic disease
* previous episode of COVID-19
* respiratory symptoms up to 14 days before the study
* history of systematic treatment with corticosteroids and/or immunosuppressant medications

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: SARSCoV2-naive adolescents with type 1 diabetes and SARSCoV2-naive healthy control adolescents who will undergo blood sampling for testing levels of antibodies against SARSCoV2 after SARSCoV2 vaccination will be consecutively included in this prospective study.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
humoral immune response after first vaccine dose | 28 days after first vaccine dose
  Levels of antibodies detected against SARSCoV2
humoral immune response after second vaccine dose | 28 days after second vaccine dose
  Levels of antibodies detected against SARSCoV2

SECONDARY OUTCOMES:
Adverse events | up to 28 days after first vaccine dose and up to 28 days after second vaccine dose
  type and number

CONTACTS AND LOCATIONS:
Overall Officials: Hamdi C Emeksiz, MD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Professor Doctor Suleyman Yalcin city Hospital, Istanbul, Eğitim Mah. Fahrettin Kerim Gökay Caddesi, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided